CLINICAL TRIAL: NCT00408616
Title: A Phase III Trial Investigating the Efficacy and Safety of Grazax in Children Aged 5-16 Years With Grass Pollen Induced Rhinoconjunctivitis With or Without Asthma
Brief Title: Efficacy and Safety of Grazax in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GT-12
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Last update posted 2009-03-09 (Estimated); Status verified 2009-03

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Grazax treatment
  Interventions: Biological: Grazax-R
- 2 (Placebo Comparator): Grazax Placebo
  Interventions: Biological: Grazax Placebo

INTERVENTIONS:
Biological: Grazax-R — Grass tablet, 75.000 SQ per day for one year
  Arms: 1
Biological: Grazax Placebo — Grazax Placebo, 0 SQ tablet per day for one year
  Arms: 2

SUMMARY:
The purpose of this study is to investigate if immunotherapy with Grazax is safe and reduces the hayfever symptoms and the use of symptom relieving medications in children during the grass pollen season

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls 5-16 years of age
* A clinical history of grass pollen induced hayfever
* Positive Skin Prick Test to Phleum pratense
* Positive specific IgE against Phleum pratense

Exclusion Criteria:

* History of seasonal hayfever symptoms (and/or asthma) caused by another allergen than Phleum pratense during or overlapping the grass pollen season
* History of perennial hayfever (and/or asthma) that needs medication due to an allergen to which the child is regularly exposed
* History of severe asthma
* Current severe atopic dermatitis

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 253 (Actual)
Dates: Start 2006-11; Primary Completion 2007-09 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Hayfever symptoms | Grass pollen season 2007
Intake of hayfever symptom relieving medication | Grass pollen season 2007

SECONDARY OUTCOMES:
Combined hayfever symptom and medication scores | Grass pollen season 2007
Asthma symptoms and medication | Grass pollen season 2007
Global Evaluation of treatment efficacy | Grass pollen season 2007
Adverse Events | 9 months
Pharmacoeconomic Assessment | 9 months
Immunological Assessment | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Friedrich Kaiser, Dr. med., Principal Investigator — Tangstedter Landstrasse 77, 22415 Hamburg, Germany
Locations (1):
- Tangstedter Landstrasse 77, Hamburg, Germany

REFERENCES:
- [Result] Bufe A, Eberle P, Franke-Beckmann E, Funck J, Kimmig M, Klimek L, Knecht R, Stephan V, Tholstrup B, Weisshaar C, Kaiser F. Safety and efficacy in children of an SQ-standardized grass allergen tablet for sublingual immunotherapy. J Allergy Clin Immunol. 2009 Jan;123(1):167-173.e7. doi: 10.1016/j.jaci.2008.10.044. PMID 19130937